CLINICAL TRIAL: NCT07079280
Title: Comparison of Acute Micro- and Macrovascular Responses to Aerobic Exercise With and Without Blood Flow Restriction in Young and Older Adults: A Randomized Crossover Trial.
Brief Title: Comparing Vascular Responses to Aerobic Exercise With and Without Blood Flow Restriction in Young and Older Adults
Acronym: UNDER PRESSURE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Egas Moniz - Cooperativa de Ensino Superior, CRL (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: UNDER PRESSURE
Record Dates: First submitted 2025-07-13; First posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Ageing; Blood Flow Restriction (BFR) Training Effects
Keywords: Aerobic Exercise; Blood Flow Restriction; Microvascular Function; Flow mediated Slowing; Arterial Stiffness; Central Blood Pressure; Young Adults; Older Adults
MeSH Terms: interventions — High-Intensity Interval Training

STUDY DESIGN:
Intervention Model Description: Parallel group crossover randomized trial
Masking Description: Outcomes will be assessed by the same experts in every time point. Participants and evaluators will be blinded until arrival of the participant for the fist experimental condition.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Aerobic Exercise with Blood Flow Restriction (Experimental)
  Interventions: Other: Low Intensity Aerobic Exercise with Blood Flow Restriction (LIAE+BFR)
- Aerobic Exercise Without Blood Flow Restriction (Active Comparator)
  Interventions: Other: High Intensity Interval Exercise (HIIE)
- No Exercise or Blood Flow Restriction (No Intervention)

INTERVENTIONS:
Other: Low Intensity Aerobic Exercise with Blood Flow Restriction (LIAE+BFR) — In the LIAE+BFR condition, participants will walk on a treadmill for 20 minutes at 30-40% of heart rate reserve (HRR), with a pneumatic cuff inflated to 1.3 times the individual's ankle systolic blood pressure, using a 5cm wide x 75cm long commercial cuff around each upper thigh.
  Treadmill speed will be adjusted dynamically to maintain target intensities, while the incline remains at 1%. Heart Rate, the Modified Borg Rate of Perceived Exertion scale, and the Rating of perceived discomfort will be continuously monitored throughout both exercise sessions to ensure adherence to the prescribed intensity levels.
  Arms: Aerobic Exercise with Blood Flow Restriction
Other: High Intensity Interval Exercise (HIIE) — In the HIIE condition, participants will perform a 20 minutes treadmill-based HIAE, alternating between 60-seconds high-intensity intervals at 60-89% HRR and 60-second active recovery intervals at 40-50% HRR.
  Treadmill speed will be adjusted dynamically to maintain target intensities, while the incline remains at 1%. Heart Rate, the Modified Borg Rate of Perceived Exertion scale, and the Rating of perceived discomfort will be continuously monitored throughout both exercise sessions to ensure adherence to the prescribed intensity levels.
  Arms: Aerobic Exercise Without Blood Flow Restriction

SUMMARY:
Aging is a major risk factor for cardiovascular disease (CVD), contributing to progressive macrovascular and microvascular dysfunction. Macrovascular impairments, such as arterial stiffening and endothelial dysfunction, reduce nitric oxide (NO) bioavailability, leading to hypertension and impaired blood flow regulation. Microvascular dysfunction exacerbates cardiovascular decline by compromising capillary perfusion and tissue oxygenation, increasing susceptibility to ischemic events. Preserving vascular function is essential for maintaining cardiovascular health in aging populations.

Low-intensity aerobic exercise (LIAE) improves cardiovascular health and mobility, particularly in populations unable to perform high-intensity exercise. However, LIAE alone often fails to induce significant vascular adaptations, such as improved arterial compliance or endothelial function, highlighting the need for optimized interventions.

Blood Flow Restriction (BFR) enhances vascular adaptations during low-intensity exercise by inducing localized hypoxia, stimulating endothelial function and arterial remodeling. While BFR may transiently increase blood pressure and arterial stiffness, its vascular benefits resemble those of high-intensity exercise at lower workloads. However, research on BFR's acute vascular effects during aerobic exercise in older adults remains limited.

Current studies have focused on perceptual and hemodynamic responses to LIAE+BFR but lack direct assessments of macrovascular (e.g., flow-mediated slowing) and microvascular function. Older adults may exhibit distinct vascular responses, yet data are scarce. This study examines acute vascular responses to LIAE+BFR and high-intensity interval exercise (HIIE) in young and older adults.

Hypothesis:

1. BFR combined with LIAE will elicit greater acute microvascular and macrovascular responses in older adults than in younger adults.
2. These responses will be comparable to HIIE without BFR, suggesting BFR enhances LIAE's efficacy to high-intensity levels.
3. Any transient vascular dysfunction (e.g., increased arterial stiffness) will normalize within 30 minutes post-exercise, supporting safety in aging populations.

DETAILED DESCRIPTION:
In this parallel-group crossover randomized trial, young and older adult participants will be randomly assigned to two experimental conditions: LIAE+BFR and HIIE. These two conditions were specifically chosen because they are known to induce similar haemodynamic responses. Each participant will visit the laboratory on three separate occasions, with at least one week between visits allowing recovery and minimizing potential carryover effects.

On Visit 1, participants will be familiarized with the exercise and testing protocols, undergo body composition measurements, and have baseline macrovascular and microvascular function evaluated twice, 30 minutes apart, in a resting condition (control). On Visits 2 and 3, participants will perform the experimental conditions in a simple randomized order, with allocation concealed until arrival at the laboratory. The simple randomization scheme sequence will be generated by Dr. XM using a web-based randomization tool (http://www.randomizer.org/) and placed in sequentially numbered, opaque, sealed envelopes to ensure allocation concealment and minimize bias. Researchers conducting field assessments will remain blinded to group allocation until the day of the first visit.

Each session will begin with 15 minutes of supine rest on a cushioned examination table, followed by baseline assessments of brachial (bSBP) and central blood pressure (cSBP), heart rate (HR), microvascular function using finger photoplethysmography (Vicorder, 80 beats medical, Berlin, Germany)., macrovascular function using FMS, and central PWV (cPWV).

After baseline assessments, participants will engage in one of the randomized aerobic exercise conditions, lasting approximately 30 minutes. The workload will be equalized considering intensity and stimulus time (intensity x duration) and the protocol is directly inspired by a previous study. In the LIAE+BFR condition, participants will walk on a treadmill (Technogym Excite Run, Technogym SpA, Cesena, Italy) for 20 minutes, using a 5 cm × 75 cm pneumatic cuff (Occlusion Cuff Pro®, Occlusion Cuff LLC, 2024) inflated to 1.3 times the individual's ankle SBP (Suga et al., 2012) The intensity will be set between 30-39% of heart rate reserve (HRR), a widely used method for prescribing aerobic exercise intensity (Liguori et al., 2021). In the HIIE condition, participants will perform a 20-minute treadmill-based high-intensity interval training, alternating between 60-seconds high-intensity intervals at 60-89% HRR and 60-second active recovery intervals at 40-50% HRR. Treadmill speed will be adjusted dynamically to maintain target intensities, while the incline remains at 1%. HR, the Modified Borg Rate of Perceived Exertion (RPE) scale, and the Rating of perceived discomfort will be continuously monitored throughout both exercise sessions to ensure adherence to the prescribed intensity levels.

Immediately after exercise, participants will return to the examination table for a 30-minute recovery period, during which brachial blood pressure, heart rate, and micro- and macrovascular function will be reassessed at 5- and 30-minutes post-exercise and compared to resting values. These post-exercise time points aim to characterize the biphasic response of macro- and microvascular function.

All participants will report to the laboratory between 8:00 AM and 12:00 PM, with room temperature controlled between 20-22°C. Participants will be instructed to avoid caffeine and alcohol for 24 hours, fully void before the session, and refrain from vigorous physical activity for 24 hours before each session, including the familiarization session.

All evaluations will be conducted by four trained physiotherapy students per participant (4:1), each with over 30 hours of training in the evaluation and exercise protocols. Throughout all sessions, a certified professional in basic life support (BLS) and automated external defibrillator (AED) use will be present at the clinic.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18-30 years and those over 60 years.

Exclusion Criteria:

* Past or current history of coronary heart disease, stroke, oncological disease, or major cardiovascular events.
* Individuals who had undergone surgery within the last two months
* Body mass index (BMI) greater than 30 kg/m²
* Declared sleep apnea
* Active kidney or liver disease
* Active tobacco smokers
* Sensory impairments
* Neurological or orthopedic functional impairments, musculoskeletal pathologies affecting exercise capacity
* Physically active for more than six months with a weekly activity level of 1,000 MET/min.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2025-10-06 (Estimated); Primary Completion 2026-05-29 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in macrovascular function | At rest and re-evaluated 5- and 30-minutes into recovery following the experimental conditions
  We will use the slowing of the pulse wave velocity (PWV) recorded between the upper arm and the wrist as an index of macrovascular function. PWV is inversely related to arterial distensibility; a widening of the brachial artery cross-section will cause a drop in post-occlusive PWV. Macrovascular function will be evaluated using EndoFMS (Vicorder, Berlin, Germany), and the response parameters are PWVmin and PWV% change from pre-occlusion values. The percentage change from initial PWV is called FMS. The default cuff placement is a 10 cm brachial cuff on the upper arm and a 7 cm wrist cuff on the selected limb. The test is performed with the patient lying horizontally, the right arm extended at a 60-degree angle, and the hand rotated palm up. After the patient relaxes, the test starts with a target occlusion pressure 30 mmHg above systolic pressure. Brachial PWV is measured between the wrist and upper arm over 10 minutes, with a 5-minute occlusion period.
Change in central arterial stiffness | At rest and re-evaluated 5- and 30-minutes into recovery following the exercise condition
  To measure arterial stiffness, we will assess carotid-femoral pulse wave velocity (cPWV) using a Vicorder module (Berlin, Germany). Participants will be in a reclined position, with a minimum of 10 minutes of rest. A 100 mm blood pressure cuff will encircle the upper thigh, and a 30 mm partial cuff will be applied around the neck at the level of the carotid arteries, above the thyroid prominence. The direct path length will be measured from the suprasternal angle to the middle of the femoral blood pressure cuff by the same operator. Both cuffs will be simultaneously inflated to 60 mm Hg to capture femoral and carotid waveforms. Continuous recordings will be obtained beat-to-beat for at least 3 minutes. Automated software will determine the wave's foot using an intersecting tangent algorithm. The time delay between the foot of the carotid and femoral waveforms will provide the average TT every 3.5 seconds.
Change in blood pressure | At rest and re-evaluated after each set and 5- and 30-minutes into recovery following the exercise condition
  The brachial artery pulse waveform obtained oscillometrically, will be analyzed using the Pulse Wave Analysis (PWA) function of the Vicorder® device (Berlin, Germany), and the aortic waveform calculated using a transfer function. This enables calculation of arterial system parameters, including cSBP, augmentation pressure (AugPress), augmentation index (AugInd), central peripheral pressure (cPP), cardiac output, and total peripheral resistance. Initial waves will be omitted, and good-quality consecutive pulse waves will be analyzed.
Change in microvascular function | At rest and re-evaluated 5- and 30-minutes into recovery following the exercise condition
  Microvascular function will be assessed using EndoCheckPAR (Vicorder, Berlin, Germany). Participants will be in a supine position with their arms comfortably positioned. Changes in the peripheral arterial dilation ratio (PAR) signal to reactive hyperemia (RH) will be measured at the fingertip with photoplethysmographs and an inflating device controlled by a computer algorithm. The RH procedure consists of a 30-second calibration, a 5-minute baseline recording, followed by 5 minutes of blood flow occlusion of the test arm using an upper arm blood pressure cuff inflated to 30 mmHg above the patient's systolic brachial pressure. After cuff deflation, the PAR tracing will be recorded for another 3 minutes. The software automatically normalizes this ratio to the concurrent signal from the contralateral, non-occluded forearm to correct for confounding variables. This ratio is then multiplied with a baseline correction factor to obtain Measured Peak, Max Reference Peak, and Max PAR.

CONTACTS AND LOCATIONS:
Locations (1):
- Egas Moniz School of Health and Science, Almada, Portugal

IPD SHARING:
Plan to Share IPD: Yes
Data obtained in this study may be provided to qualified researchers with academic interest in vascular responses to aerobic training with blood flow restriction. Data or samples shared will be coded, with no PHI included. Approval of the request and execution of all applicable agreements (i.e. a material transfer agreement) are prerequisites to the sharing of data with the requesting party.
Supporting Information: Study Protocol
Time Frame: Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis.
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information or to submit a request, please contact xmelo@egasmoniz.edu.pt

REFERENCES:
- [Background] Zhang Y, Chai S, Dai H, Chen X, Meng Z, Ying X. Vascular endothelial function and its response to moderate-intensity aerobic exercise in trained and untrained healthy young men. Sci Rep. 2024 Sep 3;14(1):20450. doi: 10.1038/s41598-024-71471-7. PMID 39242762
- [Background] Thomas HJ, Scott BR, Peiffer JJ. Acute physiological responses to low-intensity blood flow restriction cycling. J Sci Med Sport. 2018 Sep;21(9):969-974. doi: 10.1016/j.jsams.2018.01.013. Epub 2018 Apr 9. PMID 29650336
- [Background] Staunton CA, May AK, Brandner CR, Warmington SA. Haemodynamics of aerobic and resistance blood flow restriction exercise in young and older adults. Eur J Appl Physiol. 2015 Nov;115(11):2293-302. doi: 10.1007/s00421-015-3213-x. Epub 2015 Jul 4. PMID 26142277
- [Background] Formiga MF, Fay R, Hutchinson S, Locandro N, Ceballos A, Lesh A, Buscheck J, Meanor J, Owens JG, Cahalin LP. EFFECT OF AEROBIC EXERCISE TRAINING WITH AND WITHOUT BLOOD FLOW RESTRICTION ON AEROBIC CAPACITY IN HEALTHY YOUNG ADULTS: A SYSTEMATIC REVIEW WITH META-ANALYSIS. Int J Sports Phys Ther. 2020 Apr;15(2):175-187. PMID 32269850
- [Background] Chua MT, Sim A, Burns SF. Acute and Chronic Effects of Blood Flow Restricted High-Intensity Interval Training: A Systematic Review. Sports Med Open. 2022 Sep 30;8(1):122. doi: 10.1186/s40798-022-00506-y. PMID 36178530
- [Background] Bai X, Soh KG, Omar Dev RD, Talib O, Xiao W, Soh KL, Ong SL, Zhao C, Galeru O, Casaru C. Aerobic Exercise Combination Intervention to Improve Physical Performance Among the Elderly: A Systematic Review. Front Physiol. 2022 Jan 4;12:798068. doi: 10.3389/fphys.2021.798068. eCollection 2021. PMID 35058805
- [Background] Barili A, Corralo VDS, Cardoso AM, Manica A, Bonadiman BDSR, Bagatini MD, Da Silva-Grigoletto ME, de Oliveira GG, De Sa CA. Acute responses of hemodynamic and oxidative stress parameters to aerobic exercise with blood flow restriction in hypertensive elderly women. Mol Biol Rep. 2018 Oct;45(5):1099-1109. doi: 10.1007/s11033-018-4261-1. Epub 2018 Jul 20. PMID 30030775
- [Background] de Queiros VS, Rolnick N, Sabag A, Wilde P, Pecanha T, Aniceto RR, Rocha RFC, Delgado DZ, de Araujo Tinoco Cabral BG, Dantas PMS. Effect of High-Intensity Interval Exercise versus Continuous Low-Intensity Aerobic Exercise with Blood Flow Restriction on Psychophysiological Responses: A Randomized Crossover Study. J Sports Sci Med. 2024 Mar 1;23(1):114-125. doi: 10.52082/jssm.2024.114. eCollection 2024 Mar. PMID 38455431